CLINICAL TRIAL: NCT01443143
Title: A Comparison of Glycemic Stability and Variability During Consumption of Usual Diet or a Commercially Available Portion-controlled Diet Among Patients With Type 2 Diabetes
Brief Title: Blood Glucose Stability and Variability on Two Diets
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nutrisystem, Inc. (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SPO-2010-02
Record Dates: First submitted 2011-09-26; First posted 2011-09-29 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Diabetes; Obesity; Glycemic; Portion-control; Commercial diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Commercial diet (Experimental): Commercially available diet program (i.e., Nutrisystem D) that includes pre-packaged low-glycemic index portion-controlled entrees and snacks that are supplemented with grocery items in accordance with a structured meal plan.
  Interventions: Other: Portion-controlled diet
- Usual Diet (No Intervention): Participants' usual consumption of food and beverages.
  Interventions: Dietary Supplement: Usual Diet

INTERVENTIONS:
Other: Portion-controlled diet — During this diet period, participants will consume portion-controlled products from the Nutrisystem-D program for three entrees and one (women) or two (men) snacks per day. These pre-packaged portion-controlled items will be supplemented with grocery additions (fruits, vegetables, and low-fat dairy items) to provide approximately 1300 (women) to 1500 (men) calories per day. The Nutrisystem-D program (i.e., provided foods plus grocery additions) provides approximately 53% of calories from carbohydrate, 22% of calories from fat (6% from saturated fat and 0% from trans fat), and 25% of calories from protein. Women and men on the program consume approximately 1800 and 2000 mg/d, respectively, of sodium, and 31 and 35 g/d, respectively, of fiber.
  Other Names: Nutrisystem D
  Arms: Commercial diet
Dietary Supplement: Usual Diet — During the usual diet period, participants will not be given any specific instructions about what they should or should not consume. Instead, they will be told to "Eat how you would normally eat if you were not in this study."
  Arms: Usual Diet

SUMMARY:
This investigation will examine the effects of consuming a structured, portion-controlled, low-glycemic index diet (commercially available as the Nutrisystem-D program) on several indicators of glycemic stability and variability among participants with type 2 diabetes. Results on the portion-controlled diet will be compared with those on participants' usual diets in a randomized cross-over trial. The investigators expect that participants will exhibit greater glycemic stability (e.g., more time in euglycemic range) and less glycemic variability (e.g., smaller mean amplitude of glycemic excursions) while consuming the Nutrisystem D program, as compared with their usual diet.

DETAILED DESCRIPTION:
This study will investigate glycemic stability and variability in response to two diets: usual diet and a commercially available portion-controlled diet. The commercially available diet will be the Nutrisystem-D program, which consists of pre-packaged meals and snacks that are supplemented with grocery items, including fruits, vegetables, and dairy items. This trial will be a randomized cross-over trial of 15 patients with type 2 diabetes (weight stable for at least 3 months prior and medication stable throughout the trial). Participants will consume each diet for a 2-week period. During each diet period, participants will wear a blinded (i.e., providing no feedback) continuous glucose monitoring (CGM) device to assess glycemic stability and variability, and will be instructed to keep a detailed record of food and beverage intake and physical activity. The two diet/assessment periods will be separated by a 1-week washout period during which no dietary instruction will be given and no outcomes will be measured. Laboratory values (HbA1c, glucose, insulin, lipid panel) and physical measures (height, weight, waist circumference, blood pressure) will be assessed at the baseline for descriptive purposes.

Primary Hypothesis: A significantly greater percentage of CGM readings will fall in the euglycemic range (71-180 mg/dl) during consumption of the Nutrisystem-D program, as compared with Usual Diet.

Secondary Hypothesis: Participants will have significantly smaller areas under the curve, mean amplitude of glycemic excurisions, mean, standard deviation, and interquartile range of glucose values, and a smaller of percentage of values in the hypo- (</= 70 mg/dl) and hyperglycemic (>180 mg/dl) ranges during consumption of the Nutrisystem-D program, as compared with Usual Diet.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes
* Body mass index (BMI) of 27 to 45 kg/m2
* Capacity to provide written informed consent
* Willing and committed to return for all clinic visits and complete all study-related procedures
* Men and women of all racial and ethnic groups are eligible for participation

Exclusion Criteria:

* Use of hypoglycemic medications (e.g., sulfonylureas, insulin)
* Food allergies or intolerances that would render adherence to the test diets unpleasant or unsafe
* Use of anticoagulant medications (e.g., warfarin)
* Pregnant or lactating
* More than a 5% weight gain or loss within the last 3 months
* More than one alcoholic drink per day
* Binge eating disorder
* Regular use of acetaminophen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Percent of time in euglycemic range | 2 weeks
  Euglycemia will be defined as a CGM reading in the range of 71-180 mg/dl, inclusive. Percent of time in the euglycemic range each day is automatically generated by the software accompanying the CGM device. Daily values will be averaged over each of the 2-week assessment periods (i.e. during consumption of Usual Diet or Nutrisystem-D program).

SECONDARY OUTCOMES:
AUC | 2 weeks
  Area under the curve (AUC) for glucose will be calculated (using the trapezoidal method) for each day of monitoring and averaged over each of the 2-week assessment periods.
MAGE | 2 weeks
  Mean amplitude of glycemic excursions(MAGE) will be calculated (using methods described by Service et al.) for each day of monitoring and averaged over each of the 2-week assessment periods
Mean glucose | 2 weeks
  Daily values for mean blood glucose will be automatically generated by the software that accompanies the CGM device. These daily values will be averaged over each of the 2-week assessment periods.
SD of glucose values | 2 weeks
  The daily standard deviation (SD) of blood glucose values will be automatically generated by the software that accompanies the CGM device. These daily values will be averaged over each of the 2-week assessment periods.
IQR of blood glucose | 2 weeks
  The daily interquartile range(IQR) of blood glucose values will be automatically generated by the software that accompanies the CGM device. These daily values will be averaged over each of the 2-week assessment periods.
Percent of time in hypoglycemic range | 2 weeks
  Daily values for percent of time in the hypoglycemic range (< 70 mg/dl) will be automatically generated by the software that accompanies the CGM device. Daily values will be averaged over each of the 2-week assessment periods.
Percent of time in hyperglycemic range | 2 weeks
  Daily values for percent of time in the hyperlycemic range (>/= 180 mg/dl) will be automatically generated by the software that accompanies the CGM device. Daily values will be averaged over each of the 2-week assessment periods.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Wadden, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Center for Weight and Eating Disorders, Philadelphia, Pennsylvania, United States